CLINICAL TRIAL: NCT03505008
Title: MIRACLE (Methotrexate Inadequate Response Patient With Rheumatoid Arthritis Treated by Adalimumab in Combination With Low-dose Methotrexate) Study
Brief Title: Evaluation of the Optimal MTX Dose as an Add-on Therapy to Adalimumab for RA Patients in Japan, South Korea and Taiwan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keio University (Other)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yuko Kaneko, Study Principal Investigator, Keio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2E7-C000-401
Record Dates: First submitted 2018-04-16; First posted 2018-04-20 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Methotrexate; Adalimumab; Autoimmune Disease; Connective Tissue Diseases; Rheumatic Disease; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases; Connective Tissue Diseases; Rheumatic Diseases | interventions — Methotrexate; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTX-Monotherapy Group (Experimental): Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the maximum tolerated dose (MTD) of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and simple disease activity index (SDAI) remission is achieved at Week 24, the MTX therapy will continue until Week 48.
  Interventions: Drug: Methotrexate
- ADA/MTX-Maximum Tolerated Dose Group (Experimental): Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the MTD of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and SDAI remission is not achieved at Week 24, Adalimumab (ADA) 40 mg will be administered subcutaneously every other week in addition to the MTX therapy until Week 48.
  Interventions: Drug: Methotrexate; Drug: Adalimumab
- ADA/MTX-Reduced Dose Group (Experimental): Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the MTD of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and SDAI remission is not achieved at Week 24, Adalimumab (ADA) 40 mg will be administered subcutaneously every other week in addition to low-dose MTX (6 to 8 mg/week) treatment until Week 48.
  Interventions: Drug: Methotrexate; Drug: Adalimumab

INTERVENTIONS:
Drug: Methotrexate — Route of Administration: Oral
  Other Names: MTX
Drug: Adalimumab — Route of Administration: Subcutaneous
  Other Names: ADA
  Arms: ADA/MTX-Maximum Tolerated Dose Group; ADA/MTX-Reduced Dose Group

SUMMARY:
This study will be conducted in Japan, South Korea and Taiwan to evaluate the optimal dosage of methotrexate (MTX) as an add-on therapy to adalimumab (ADA) in participants with rheumatoid arthritis (RA) who have not achieved remission by MTX monotherapy.

DETAILED DESCRIPTION:
The erythrocyte MTX-polyglutamates (MTX-PG) concentration will be measured to evaluate its relationship to the efficacy and safety of MTX therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years (≥20 years in Taiwan) at the time of informed consent
2. Patients who meet the 1987 revised ACR criteria or 2010 ACR/EULAR criteria
3. Patients who have RA within 2 years from initial diagnosis to informed consent
4. Patients who were previously untreated with MTX, JAK inhibitor, or bDMARDs
5. Patients who have disease activity of SDAI >11 at screening
6. Patients who are no need for concomitant use of DMARDs other than hydroxychloroquine (only in South Korea and Taiwan) and study drugs during the study as judged by principal investigator/sub-investigator at screening
7. Patients who are no need for concomitant use of corticoid steroid equivalent to >10 mg/day prednisolone during the study as judged by principal investigator/sub-investigator at screening.
8. Female of child-bearing potential who can use appropriate contraceptive during the study, female in whom time from menopause to informed consent is ≥1 year, or female of no child-bearing potential through sterilization (bilateral tubal ligation, bilateral ovariectomy or hysterectomy, etc.)
9. Virile male who can use appropriate contraceptive during the study
10. Patients who can adequately understand this study procedures, and voluntarily consent in writing to take part in this study (consent of a legally-acceptable representative is also required for patients aged <20 years in Japan and aged <19 years in South Korea)

Exclusion Criteria:

1. Patients who currently have a malignant tumor, except for non-melanoma forms of skin cancer limited within epidermis, and uterine cervix cancer limited within epidermis
2. Patients who have serious infections such as sepsis
3. Patients who have active tuberculosis
4. Patients who have a history or current complication of demyelinating disease such as multiple sclerosis
5. Patients who have congestive heart failure
6. Pregnant female, or female who intend to conceive during the study period
7. Patients who have bone marrow depression and whom investigator considered ineligible
8. Patients who have chronic liver disease and whom investigator considered ineligible, and who is positive for HBs antigen
9. Patients who have nephropathy and whom investigator considered ineligible
10. Lactating female
11. Patients who have pleural effusion or ascites
12. Patients with a known hypersensitivity to MTX or ADA
13. Patients otherwise whom principal investigator/sub-investigator considered medically ineligible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Kaneko, MD, PhD, Principal Investigator — Division of Rheumatology, Department of Internal Medicine, Keio University School of Medicine
Locations (24):
- Japan (12):
  - Fujita Health University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - Hiroshima University Hospital, Hiroshima
  - Kawasaki Municipal Hospital, Kanagawa
  - Tokai University Hospital, Kanagawa
  - Tohoku University Hospital, Miyagi
  - Nagoya University Hospital, Nagoya
  - Seirei Hamamatsu General Hospital, Shizuoka
  - Keio University Hospital, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Toho University Ohashi Medical Center, Tokyo
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (6):
  - Chang Gung Medical Foundation, Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation, Linkou Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- [Derived] Tamai H, Ikeda K, Miyamoto T, Taguchi H, Kuo CF, Shin K, Hirata S, Okano Y, Sato S, Yasuoka H, Kuwana M, Ishii T, Kameda H, Kojima T, Nishi Y, Mori M, Miyagishi H, Toshima G, Sato Y, Tsai WC, Takeuchi T, Kaneko Y; MIRACLE Study Group. Association of methotrexate polyglutamates concentration with methotrexate efficacy and safety in patients with rheumatoid arthritis treated with predefined dose: results from the MIRACLE trial. Ann Rheum Dis. 2025 Jan;84(1):41-48. doi: 10.1136/ard-2024-226350. Epub 2025 Jan 2. PMID 39874232
- [Derived] Tamai H, Ikeda K, Miyamoto T, Taguchi H, Kuo CF, Shin K, Hirata S, Okano Y, Sato S, Yasuoka H, Kuwana M, Ishii T, Kameda H, Kojima T, Taninaga T, Mori M, Miyagishi H, Sato Y, Tsai WC, Takeuchi T, Kaneko Y; MIRACLE study collaborators. Reduced versus maximum tolerated methotrexate dose concomitant with adalimumab in patients with rheumatoid arthritis (MIRACLE): a randomised, open-label, non-inferiority trial. Lancet Rheumatol. 2023 Apr;5(4):e215-e224. doi: 10.1016/S2665-9913(23)00070-X. PMID 38251524

RESULTS

PARTICIPANT FLOW:
Groups:
- MTX-Monotherapy Before Week 24 Randomization: Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the maximum tolerated dose (MTD) of ≤25 mg/week up to Week 12, and maintained until Week 24.
  Methotrexate: Route of Administration: Oral
- MTX-Monotherapy Group After Week 24: Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the maximum tolerated dose (MTD) of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and simple disease activity index (SDAI) remission is achieved at Week 24, the MTX therapy will continue until Week 48.
  Methotrexate: Route of Administration: Oral
- ADA/MTX-Maximum Tolerated Dose Group After Week 24: Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the MTD of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and SDAI remission is not achieved at Week 24, Adalimumab (ADA) 40 mg will be administered subcutaneously every other week in addition to the MTX therapy until Week 48.
  Methotrexate: Route of Administration: Oral
  Adalimumab: Route of Administration: Subcutaneous
- ADA/MTX-Reduced Dose Group After Week 24: Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the MTD of ≤25 mg/week up to Week 12, and maintained until Week 24. If the dosage of MTX is maintained ≥ 10 mg/week and SDAI remission is not achieved at Week 24, Adalimumab (ADA) 40 mg will be administered subcutaneously every other week in addition to low-dose MTX (6 to 8 mg/week) treatment until Week 48.
  Methotrexate: Route of Administration: Oral
  Adalimumab: Route of Administration: Subcutaneous
Period: Before Week 24 Randomization
Arm/Group | MTX-Monotherapy Before Week 24 Randomization | MTX-Monotherapy Group After Week 24 | ADA/MTX-Maximum Tolerated Dose Group After Week 24 | ADA/MTX-Reduced Dose Group After Week 24
Started (FAS at week 0) | 291 | 0 | 0 | 0
Completed (FAS at week 24) | 239 | 0 | 0 | 0
Not Completed | 52 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 24 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 0 | 0 | 0
Not completed — Methotrexate <10 mg/week at Week 24 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Inadequate Methotrexate Adherence | 1 | 0 | 0 | 0
Not completed — Complication | 1 | 0 | 0 | 0
Period: After Week 24 Randomization
Arm/Group | MTX-Monotherapy Before Week 24 Randomization | MTX-Monotherapy Group After Week 24 | ADA/MTX-Maximum Tolerated Dose Group After Week 24 | ADA/MTX-Reduced Dose Group After Week 24
Started (FAS at week 24. Participants who achieved SDAI remission at Week 24 were allocated to MTX-Monotherapy Group. Only participants who did not achieve SDAI remission at Week 24 were randomized and received Adalimumab in addition to the MTX therapy.) | 0 | 105 | 68 | 66
Completed (FAS at week 48) | 0 | 101 | 59 | 58
Not Completed | 0 | 4 | 9 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Lack of Efficacy | 0 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Full-analysis Set: Participants will receive Methotrexate (MTX) at a starting dose of 6 to 8 mg/week, which will be promptly escalated to the maximum tolerated dose (MTD) of ≤25 mg/week up to Week 12, and maintained until Week 24.
  Methotrexate: Route of Administration: Oral
Arm/Group | Full-analysis Set
Number analyzed (Participants) | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217
  Male | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 290
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 194
  South Korea | 55
  Taiwan | 42
Duration from the Diagnosis of Rheumatoid Arthritis [Mean (Standard Deviation); unit: days] | 21.1 (56.2)
Bodyweight [Mean (Standard Deviation); unit: kg] | 58.2 (11.4)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m²] | 82.0 (20.2)
Current or Past Smoker [Count of Participants; unit: Participants] | 102
Simplified Disease Activity Index (SDAI) [Mean (Standard Deviation); unit: scores on a scale] — SDAI is a validated combined index of rheumatoid arthritis disease activity, defined as the sum of Swollen Joint Count (0-28), Tender Joint Count (0-28), Patient's Global Assessment of Disease Activity (range of 0 [none] to 10 [most severe]), Physician's Global Assessment of Disease Activity (range of 0 [none] to 10 [most severe]), and C-reactive protein (mg/dL, 0- with no maximum limit).
  Higher scores represent higher disease activity. SDAI ≤ 3.3 indicates disease remission, > 3.3 to 11 = low disease activity, > 11 to 26 = moderate disease activity, and > 26 = high disease activity.
  scores on a scale | 26.5 (12.4)
28-Joint Disease Activity Score of Erythrocyte Sedimentation Rate (DAS28-ESR) [Mean (Standard Deviation); unit: scores on a scale] — DAS28-ESR is a validated combined index of rheumatoid arthritis disease activity calculated as 0.56*√(Tender Joint Count, 0-28) + 0.28*√(Swollen Joint Count, 0-28) + 0.7*ln(Erythrocyte Sedimentation Rate, mm/hr) + 0.014*(Patient's global assessment, 0-100 mm on visual analogue scale).
  Scores on the DAS28-ESR range from 0 to 10, where higher scores represent higher disease activity.
  DAS28-ESR < 2.6 indicates disease remission, ≥ 2.6 to 3.2 = low disease activity, > 3.2 to 5.1 = moderate disease activity, and > 5.1 = high disease activity.
  scores on a scale | 5.2 (1.1)
Health Assessment Questionnaire - Disability Index (HAQ-DI) [Mean (Standard Deviation); unit: scores on a scale] — HAQ-DI is a patient-reported questionnaire, consists of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week as: without any difficulty (0); with some difficulty (1); with much difficulty (2); unable to do (3). Scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0=no disability and 3=very severe, high-dependency disability. Normal physical function is defined by HAQ-DI score of < 0.5.
  scores on a scale | 0.9 (0.7)
Rheumatoid Factor Positive [Count of Participants; unit: Participants] — Population: One person was not tested.
  Participants
    number analyzed (Participants) | 290
    (all) | 213
Anti-cyclic Citrullinated Peptide Antibody Positive [Count of Participants; unit: Participants] — Population: Two people were not tested.
  Participants
    number analyzed (Participants) | 289
    (all) | 211
Comorbidities [Count of Participants; unit: Participants] | 127

OUTCOME MEASURES:

1. Primary Outcome: Simple Disease Activity Index (SDAI) Remission Rate at Week 48 in mFAS
Description: SDAI is a validated combined index of rheumatoid arthritis disease activity, defined as the sum of Swollen Joint Count (0-28), Tender Joint Count (0-28), Patient's Global Assessment of Disease Activity (measured on a visual analogue scale with a range of 0 [none] to 10 [most severe]), Physician's Global Assessment of Disease Activity (measured on a visual analogue scale with a range of 0 [none] to 10 [most severe]), and C-reactive protein (mg/dL).
  Higher scores represent higher disease activity. SDAI ≤ 3.3 indicates disease remission, > 3.4 to 11 = low disease activity, > 11 to 26 = moderate disease activity, and > 26 = high disease activity.
Time Frame: Week 48
Population: In the modified Full Analysis Set based on non-responder imputation. The modified Full Analysis Set was defined as those with evaluable data set at one or more timepoints after randomization including 66 of 68 subjects in ADA/MTX-Maximum Tolerated Dose Group and 61 of 66 subjects in ADA/MTX-Reduced Dose Group.
  Primary and secondary analysis were performed in subjects randomized at week 24 and planed to receive ADA, not including MTX-Monotherapy Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 66 | 61
Participants | 25 | 27
Statistical Analysis 1: Comparison: ADA/MTX-Maximum Tolerated Dose Group vs ADA/MTX-Reduced Dose Group; Test type: Non-Inferiority — Two-sided 90% CI for the intergroup difference in SDAI remission rates to exceed the non-inferiority margin of -15%; Risk Difference (RD) = 0

2. Secondary Outcome: Simple Disease Activity Index (SDAI) Remission Rate at Week 48 in PPS
Description: as for outcome 1
Time Frame: Week 48
Population: In the Per Protocol Set based on non-responder imputation. The Per Protocol Set is defined as a group of subjects among modified Full Analysis Set who adequately complied with the protocol including 58 of 66 subjects in ADA/MTX-Maximum Tolerated Dose Group and 61 of 61 subjects in ADA/MTX-Reduced Dose Group.
  Primary and secondary analysis were performed in subjects randomized at week 24 and planed to receive ADA, not including MTX-Monotherapy Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 58 | 61
Participants | 23 | 27

3. Secondary Outcome: American College of Rheumatology (ACR) 20 Response Rate at Week 48
Description: ACR 20 response is defined as a subject meeting all of the following 3 criteria based on the evaluation results of tender joint count, swollen joint count, VAS (physician- and patient reported), HAQ, and CRP. Also, the proportion of ACR 20 response will be referred to as ACR 20 response rate.
  * ≥20% improvement in the tender joint count (of the total 68 joints) compared to Week 0 of treatment
  * ≥20% improvement in the swollen joint count (of the total 66 joints) compared to Week 0 of treatment
  * ≥20% improvement in ≥3 of 5 parameters (physician- and patient-reported disease activities, patient-reported pain score, HAQ, and CRP) compared to Week 0 of treatment
Time Frame: Week 48
Population: In the Full Analysis Set based on non-responder imputation. Primary and secondary analysis were performed in subjects randomized at week 24 and planed to receive ADA, not including MTX-Monotherapy Group.
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 68 | 66
Participants | 47 | 47

4. Secondary Outcome: American College of Rheumatology (ACR) 50 Response Rate at Week 48
Description: ACR 50 response is defined as a subject meeting all of the following 3 criteria based on the evaluation results of tender joint count, swollen joint count, VAS (physician- and patient reported), HAQ, and CRP. Also, the proportion of ACR 50 response will be referred to as ACR 50 response rate.
  * ≥50% improvement in the tender joint count (of the total 68 joints) compared to Week 0 of treatment
  * ≥50% improvement in the swollen joint count (of the total 66 joints) compared to Week 0 of treatment
  * ≥50% improvement in ≥3 of 5 parameters (physician- and patient-reported disease activities, patient-reported pain score, HAQ, and CRP) compared to Week 0 of treatment
Time Frame: Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 68 | 66
Participants | 36 | 38

5. Secondary Outcome: American College of Rheumatology (ACR) 70 Response Rate at Week 48
Description: ACR 70 response is defined as a subject meeting all of the following 3 criteria based on the evaluation results of tender joint count, swollen joint count, VAS (physician- and patient reported), HAQ, and CRP. Also, the proportion of ACR 70 response will be referred to as ACR 70 response rate.
  * ≥70% improvement in the tender joint count (of the total 68 joints) compared to Week 0 of treatment
  * ≥70% improvement in the swollen joint count (of the total 66 joints) compared to Week 0 of treatment
  * ≥70% improvement in ≥3 of 5 parameters (physician- and patient-reported disease activities, patient-reported pain score, HAQ, and CRP) compared to Week 0 of treatment
Time Frame: Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 68 | 66
Participants | 22 | 26

6. Secondary Outcome: Health Assessment Questionnaire - Disability Index ≤0.5 at Week 48
Description: HAQ-DI is a patient-reported questionnaire, consists of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week as: without any difficulty (0); with some difficulty (1); with much difficulty (2); unable to do (3). Scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0=no disability and 3=very severe, high-dependency disability. Normal physical function is defined by HAQ-DI score of < 0.5.
Time Frame: Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 68 | 66
Participants | 40 | 41

7. Secondary Outcome: Change in Modified Total Sharp Score ≤ 0.5 at Week 48
Description: Bone erosions will be evaluated for each region from a scale of 0 (no damage) to 5 (complete collapse of the joint). The score will be 0 to 5 for each hand joint, and 0 to 10 for each foot joint. The maximum total erosion score of both hands will be 160 points, and that of both feet will be 120 points.
  Joint space narrowing will be evaluated for each region from a scale of 0 (no damage) to 4 (ankylosis or luxation). The maximum total joint space narrowing score of both hands will be 120 points, and that of both feet will be 48 points.
  Erosion scores and joint space narrowing scores were added to obtain the mTSS (range from 0 to 448).
Time Frame: Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADA/MTX-Maximum Tolerated Dose Group | ADA/MTX-Reduced Dose Group
Number analyzed (Participants) | 68 | 66
Participants | 45 | 41

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: All adverse events were followed up for 70 days from the final dose of study drug or until recovery, whichever comes first.
Groups:
- All From Week 0 to Week 48: Participants in Safety Analysis Set
Arm/Group | All From Week 0 to Week 48 | MTX-Monotherapy Before Week 24 Randomization | MTX-Monotherapy Group After Week 24 | ADA/MTX-Maximum Tolerated Dose Group After Week 24 | ADA/MTX-Reduced Dose Group After Week 24
All-Cause Mortality (participants affected / at risk) | 0/291 | 0/291 | 0/105 | 0/68 | 0/66
Serious Adverse Events (participants affected / at risk) | 23/291 | 9/291 | 6/105 | 5/68 | 3/66
Other Adverse Events (participants affected / at risk) | 122/291 | 94/291 | 25/105 | 14/68 | 6/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All From Week 0 to Week 48 (N=291) | MTX-Monotherapy Before Week 24 Randomization (N=291) | MTX-Monotherapy Group After Week 24 (N=105) | ADA/MTX-Maximum Tolerated Dose Group After Week 24 (N=68) | ADA/MTX-Reduced Dose Group After Week 24 (N=66)
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All From Week 0 to Week 48 (N=291) | MTX-Monotherapy Before Week 24 Randomization (N=291) | MTX-Monotherapy Group After Week 24 (N=105) | ADA/MTX-Maximum Tolerated Dose Group After Week 24 (N=68) | ADA/MTX-Reduced Dose Group After Week 24 (N=66)
Liver function test abnormal (Investigations) | 37 | 24 | 8 | 6 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 13 | 5 | 0 | 0
Nasopharyngitis (Infections and infestations) | 17 | 13 | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 16 | 14 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 13 | 9 | 6 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 5 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 4 | 2 | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 4 | 4 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 3 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 3 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 0 | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 3 | 0 | 0 | 0
Transaminases increased (Investigations) | 3 | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/08/NCT03505008/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT03505008/SAP_001.pdf